CLINICAL TRIAL: NCT05303415
Title: Study of Low-intensity Focused Ultrasound Effects on Heat Evoked fMRI Signals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-247
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LIFU, heat evoked fMRI signals (Experimental): fMRI resting and heat evoked signals performed after LIFU application to known brain region of interest or active sham region (within participant all conditions tested).
  Interventions: Other: Neuromodulation with low-intensity focused ultrasound

INTERVENTIONS:
Other: Neuromodulation with low-intensity focused ultrasound — Application of LIFU to induce temporary neuromodulation, effects tested with resting state and heat evoked (QST) fMRI signals

SUMMARY:
Study aims to examine the effects of noninvasive brain stimulation on brain signals. This insight may have potential clinical implications for addiction, pain, and mental health populations. Participants will receive MRI and CT imaging. Participants receive low-intensity focused ultrasound (LIFU) to temporarily change brain activity. Participants then receive fMRI scans to measure changes in both resting and heat evoked brain signaling using a quantitative sensory testing device. Heart rate, blood pressure, respiratory rate, and skin moisture is monitored. Participants complete a battery of questionnaires, both behavioral and symptom monitoring. The study takes place over 4 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, all ethnicities, who understand and speak English.

Exclusion Criteria:

Claustrophobia (scanning environment may be uncomfortable). Contraindications to MRI: including pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.

Contraindications to CT: pregnancy Active medical disorder or treatment with potential CNS effects (e.g. Alzheimer's) History of neurologic disorder. (e.g. Parkinson's, Epilepsy, or Essential Tremor) History of head injury resulting in loss of consciousness for >10 minutes. History of alcohol or drug dependence (through self-report).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
fMRI BOLD Signals | Participant study duration, approximately 3 weeks.
  Changes in fMRI BOLD signal

SECONDARY OUTCOMES:
Changes in self-reported perceived pain | Participant study duration, approximately 3 weeks.
  Change in subject perceived pain rating report on a numerical rating scale (0-10, 0 no pain, 10 worst pain)

OTHER OUTCOMES:
Monitoring changes to physiological measures | Participant study duration, approximately 3 weeks.
  Monitoring for any changes to heartrate, blood pressure, respiratory rate, or galvanic skin response.

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No